CLINICAL TRIAL: NCT01001546
Title: Internet-Based Smoking Cessation for OEF/OIF Veterans
Brief Title: Internet-Based Smoking Cessation for Operations Enduring Freedom and Iraqi Freedom (OEF/OIF) Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 08-032
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-12

CONDITIONS: Smoking Cessation
Keywords: Veterans; Smoking cessation; Operation Enduring Freedom; Operation Iraqi Freedom
MeSH Terms: conditions — Smoking Cessation | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Internet-based smoking cessation
  Interventions: Behavioral: Internet-based
- Arm 2 (Other): Clinic-based smoking cessation
  Interventions: Behavioral: Standard Clinic-Based

INTERVENTIONS:
Behavioral: Internet-based — Veterans randomized to the QuitNet will immediately be given access to the Premium, lifetime membership services.
  Other Names: Intervention
  Arms: Arm 1
Behavioral: Standard Clinic-Based — Veterans randomized to the control condition will have a consult placed to the Durham VA Medical Center (DVAMC) specialty Smoking Cessation Clinic placed on their behalf.
  Other Names: Control
  Arms: Arm 2

SUMMARY:
The overarching aim of the study is to evaluate in a randomized trial the impact of an internet intervention compared to a standard clinic-based control group to promote smoking cessation among Operation Enduring Freedom and Operation Iraqi Freedom (OEF/OIF) veterans.

DETAILED DESCRIPTION:
Project Background: Veterans returning from Iraq and Afghanistan are smoking at high rates and are at elevated risk for the development of smoking related illness. Intensive speciality clinic-based tobacco cessation programs have high efficacy, are more cost effective than less intensive approaches, and are employed by most VA medical centers. These programs, however, are infrequently attended by veterans, limiting the impact on prevalence, disease burden, and economic costs of smoking. An internet-based smoking cessation intervention could be an effective, low-cost method to implement evidence based smoking cessation principles. The internet could significantly increase the impact of smoking cessation efforts over current approaches by avoiding barriers that limit utilization of existing clinic-based services.

Project Objectives: The goal of the study is to evaluate the impact of an internet-based intervention in comparison to standard VA speciality clinic-based care in promoting smoking cessation in returning veterans. Accordingly, the specific aims and hypotheses are:

AIM 1: To evaluate the impact of an internet-based smoking cessation intervention on rates of abstinence from cigarettes (self-reported 7-day point prevalent abstinence) at 3 months and 12-month post-treatment follow-ups.

Hypothesis 1: Abstinence rates will be significantly higher among veterans randomized to the web-based intervention than those randomized to VA specialty cessation care.

AIM 2: To evaluate the impact of an internet-based smoking cessation intervention on reach of smoking cessation treatment.

Hypothesis 2.1: Internet-based treatment will result in increased reach as measured by the proportion of patients who access care. Hypothesis 2.2: Internet-based treatment will result in engagement in treatment as measured by the proportion of patients that make at least one quit attempt.

AIM 3: To evaluate the relative cost-effectiveness of the standard specialty care intervention to the web-based intervention.

Project Methods: Proposed is a trial in which 410 OEF/OIF veteran smokers will be randomized to receive either an internet-based smoking cessation intervention and nicotine replacement therapy or referral to VA specialty smoking cessation care, which includes behavioral therapy, group counseling, telephone counseling, self-help materials, and choice of smoking cessation aid (pharmacotherapy).

Participating patients will be surveyed at 3 months post-intervention and at 12 months. The primary outcome of the trial is a 7-day point prevalence abstinence at the 3-month post intervention follow-up, as measured by self-report and verified by cotinine assay.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in DVAMC for ongoing care
* Served during OEF/OIF
* Current smokers willing to make a quit attempt in the next 30 days

Exclusion Criteria:

* Active diagnosis of psychosis in the medical record
* Diagnosis of severe dementia in the medical record
* Does not have access to a telephone
* Severely impaired hearing or speech (veterans must be able to respond to phone calls)
* Refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2010-05; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S. Calhoun, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Gierisch JM, Bastian LA, Calhoun PS, McDuffie JR, Williams JW Jr. Smoking cessation interventions for patients with depression: a systematic review and meta-analysis. J Gen Intern Med. 2012 Mar;27(3):351-60. doi: 10.1007/s11606-011-1915-2. Epub 2011 Oct 26. PMID 22038468
- [Result] Zaborowski DE, Dedert EA, Straits-Troster K, Lee S, Wilson SM, Calhoun PS, Moore SD, Acheson S, Hamlett-Berry KW, Beckham JC. Public health clinical demonstration project for smoking cessation in american veterans who served since september 11, 2001. J Addict Med. 2011 Mar;5(1):79-83. doi: 10.1097/ADM.0b013e3181df97d5. PMID 21769051
- [Result] Calhoun PS, Levin HF, Dedert EA, Johnson Y; VA Mid-Atlantic Mental Illness Research, Education, Clinical Center Registry Workgroup; Beckham JC. The relationship between posttraumatic stress disorder and smoking outcome expectancies among U.S. military veterans who served since September 11, 2001. J Trauma Stress. 2011 Jun;24(3):303-8. doi: 10.1002/jts.20634. Epub 2011 Apr 26. PMID 21523829
- [Result] Straits-Troster K, Acheson S, Beckham JC, Calhoun PS, Gierisch JM, Hamlett-Berry K. Tobacco use and cessation among returning combat veterans: A mixed methods study. [Abstract]. Behavioral medicine update : a publication of the Society of Behavioral Medicine. 2010 Apr 10; 39(S1).
- [Result] Gierisch JM, Straits-Troster K, Calhoun PS, Beckham JC, Acheson S, Hamlett-Berry K. Tobacco use among Iraq- and Afghanistan-era veterans: a qualitative study of barriers, facilitators, and treatment preferences. Prev Chronic Dis. 2012;9:E58. doi: 10.5888/pcd9.110131. Epub 2012 Feb 16. PMID 22338598

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Internet-based smoking cessation
  Internet-based: Veterans randomized to the QuitNet will immediately be given access to the Premium, lifetime membership services.
- Control: Clinic-based smoking cessation
  Standard Clinic-Based: Veterans randomized to the control condition will have a consult placed to the DVAMC specialty Smoking Cessation Clinic placed on their behalf.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 206 | 207
Completed | 206 | 207
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 206 | 207 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (13.7) | 42.9 (14.4) | 43.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 175 | 174 | 349
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 194 | 199 | 393
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 7 | 10
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 76 | 86 | 162
  White | 105 | 104 | 209
  More than one race | 19 | 9 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 206 | 207 | 413

OUTCOME MEASURES:

1. Primary Outcome: The Impact of an Internet Intervention on Rates of Abstinence From Cigarettes (Self-reported 7-day Point Prevalent Abstinence)
Time Frame: 3 months post treatment
Measure: Number; unit: percentage of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 206 | 207
percentage of participants | 34.4 | 24.7

ADVERSE EVENTS:
Time Frame: The reporting period for adverse events was the duration of study participation for each participant:12 months from the date of enrollment.
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 9/206 | 7/207
Other Adverse Events (participants affected / at risk) | 9/206 | 8/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=206) | Control (N=207)
Hospitalization - mental health (Psychiatric disorders) | 1 (1) | 3 (3)
Hospitalization - respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hospitalization - cardiac (Cardiac disorders) | 2 (2) | 0 (0)
Hospitalization - knee surgery (Surgical and medical procedures) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=206) | Control (N=207)
Adverse reaction to Nicotine Replacement Medication (NRT) (Gastrointestinal disorders) | 3 (3) | 2 (2)
Motor Vehicle Accident (Social circumstances) | 0 (0) | 2 (2) — Not seriously injured
Adverse reaction to Nicotine Replacement Medication (NRT) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Adverse reaction to Nicotine Replacement Medication (NRT) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pregnancy/Childbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Minor Procedure (Surgical and medical procedures) | 1 (1) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes